CLINICAL TRIAL: NCT01689064
Title: Comparison of the Posterior Septectomy and Stamm Approach to Endoscopic Pituitary Adenoma Resection: A Randomized, Single-blind Trial
Brief Title: Comparison of Surgical Approach to Endoscopic Pituitary Adenoma Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Luke Rudmik, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-24588
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Pituitary Adenoma; Posterior Septectomy; Stamm Approach; Quality of Life
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posterior Septectomy (Active Comparator): Patient will be randomized to a study arm. The patient will be blinded to the approach. The surgeon will have performed at least 10 procedures previous for each approach. The surgeon will maintain the following surgical practives: preservation of both middle turbinates, preservation of one superior turbinate (to minimize olfactory injury), elevation of a nasoseptal flap, the use of a combination of gelform, surgicel and nasapore dissolvable spacer placed within the surgical defect. These practices are all standard of care. Patient will start Neilmed high volume low pressure saline irrigation three times daily starting on post operative day five. Patients will receive prophylactic antibiotics for fourteen days post operatively.
  Interventions: Procedure: Posterior Septectomy
- Stamm Approach (Experimental): Patient will be randomized a study arm. The patient will be blinded to the approach. The surgeon will have performed at least 10 procedures previous for each approach. The surgeon will maintain the following surgical practives: preservation of both middle turbinates, preservation of one superior turbinate (to minimize olfactory injury), elevation of a nasoseptal flap, the use of a combination of gelform, surgicel and nasapore dissolvable spacer placed within the surgical defect. These practices are all standard of care. Patient will start Neilmed high volume low pressure saline irrigation three times daily starting on post operative day five. Patients will receive prophylactic antibiotics for fourteen days post operatively.
  Interventions: Procedure: Stamm Approach

INTERVENTIONS:
Procedure: Stamm Approach
  Arms: Stamm Approach
Procedure: Posterior Septectomy
  Arms: Posterior Septectomy

SUMMARY:
The purpose of this study is to determine if there is a significant difference in sinonasal disease specific quality of life and utility scores between patients undergoing the posterior septectomy or Stamm approach during endoscopic pituitary adenoma resection.

DETAILED DESCRIPTION:
Pituitary adenoma's represent 10 to 25% of all central nervous system (CNS) neoplasms and have an estimated population prevalence of 94 per 100,000. Asymptomatic adenomas go largely undetected since there is no screening protocol implemented with the purpose for early identification. Asymptomatic adenomas can be detected incidentally on CNS imaging for other indications in approximately 10% of studies and rarely require surgical intervention. In 2011, the Endocrine Society published practice guidelines on the management of pituitary incidentalomas and provided the surgical indications. Incidental microadenoma's (< 10 mm) rarely need surgical intervention, however, incidental macroadenoma's (> 10 mm) often required surgical resection due to the proximity of the optic nerves and chiasm.

Most symptomatic pituitary adenomas require transnasal transsphenoid surgical resection. Due to the potential for hormone secretion and location to vital structures such as the optic chiasm/nerves, carotid artery, and cavernous sinus, management of symptomatic pituitary adenomas often require a multi-disciplinary team involving neurosurgery, otolaryngology, neuroophthalmology, and endocrinology. Traditionally the microscope was used for visualization during pituitary tumor surgery, however with recent technologic advances, the endoscopic approach has largely replaced the microscopic approach. A recent systematic review and meta-analysis compared the microscopic and endoscopic approaches and have demonstrated that the endoscopic approach results in a significant reduction in the rate of cerebral spinal fluid (CSF) leak, improved tumor resection, improved patient comfort, and reduced hospital length of stay. Furthermore, the endoscopic approach appears to provide an overall cost savings compared to the microscopic approach.

Several recent studies have demonstrated that the endoscopic approach for pituitary adenoma resection results in improved disease-specific quality of life (QoL) and general QoL. All studies have utilized the posterior septectomy approach which involves removing the posterior nasal septum to create a common posterior nasal cavity. The open posterior nasal cavity provides excellent surgical access to the sphenoid sinus and pituitary gland. Disadvantages of the posterior septectomy approach include the permanent posterior septal perforation which may predispose to postoperative crusting and epistaxis. A recent article by Stamm et al. described a novel endoscopic approach whereby the posterior septal mucosa is preserved while still providing excellent access to the sphenoid. The primary advantage of this approach is preventing a posterior septal defect, however disadvantages include being a more challenging technique and the potential for reduced surgical visualization. Furthermore, there is still a risk of a septal perforation due to intraoperative trauma and significant postoperative crusting which often develops along the surface of the healing septal mucosa. Both endoscopic approaches have inherent advantages and disadvantages and there has been no study comparing these approaches. Surgeons performing endoscopic pituitary tumor resections utilize both approaches and neither is considered the standard of care.

The purpose of this randomized, single-blinded study is to determine the clinical outcomes between the posterior septectomy and Stamm approach for endoscopic pituitary adenoma resection. We hypothesize that there will be no difference in disease-specific QoL and general QoL between the two surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Diagnosis of a pituitary adenoma requiring resection defined as pituitary lesion with any of the following:

  1. Neuroimaging or clinical evidence of apoplexy
  2. Decline in central visual acuity worse than (best-corrected) Snellen equivalent of 20/25 in either eye
  3. clinically significant visual field loss as determined by Humphrey or Goldmann perimetry
  4. Clinically significant cranial nerve deficit
  5. Clinically relevant neuroendocrine deficit
  6. Intolerance of optimal medical management
* Patient electing endoscopic resection approach

Exclusion Criteria:

* Concurrent chronic rhinosinusitis
* Revision pituitary adenoma resections
* Severe medical co-morbidities with the inability to undergo general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | Pre-operative and Post-operative (2 weeks, 6 weeks, 3 months and 6 months)
  To determine the change in quality of life scores between the two groups at 2 weeks, 6 weeks, 3 months and 6 months using the anterior skull base nasal inventory questionnaire, the SinoNasal outcome test-22 questionnaire and the EQ-5D questionnaire.

SECONDARY OUTCOMES:
Change in Symptom Score | Pre-operative and Post-operative (2 weeks, 6 weeks, 3 months and 6 months)
  To determine the change in symptom score between the two groups at 2 weeks, 6 weeks, 3 months and 6 months using the VAS Nasal Symptom score.
Change in Utility Score | Pre-operative and Post-operative (2 weeks, 6 weeks, 3 months and 6 months)
  To determine the change in utility score between the two groups at 2 weeks, 6 weeks, 3 months and 6 months.
Change in Endoscopic Sinus Score | Pre-operative and Post-operative (2 weeks, 6 weeks, 3 months and 6 months)
  To determine the change in endoscopic sinus score between the two groups at 2 weeks, 6 weeks, 3 months and 6 months using the endoscopic grading - Using both the Lund-Kennedy and POSE endoscopic scoring system.
Change in Olfaction | Pre-operative and Post-operative (6 months)
  To determine the change in olfaction between the two groups at 6 months using the Smell Identification Test (SIT).

CONTACTS AND LOCATIONS:
Overall Officials: Luke Rudmik, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Daly AF, Rixhon M, Adam C, Dempegioti A, Tichomirowa MA, Beckers A. High prevalence of pituitary adenomas: a cross-sectional study in the province of Liege, Belgium. J Clin Endocrinol Metab. 2006 Dec;91(12):4769-75. doi: 10.1210/jc.2006-1668. Epub 2006 Sep 12. PMID 16968795
- [Background] Hall WA, Luciano MG, Doppman JL, Patronas NJ, Oldfield EH. Pituitary magnetic resonance imaging in normal human volunteers: occult adenomas in the general population. Ann Intern Med. 1994 May 15;120(10):817-20. doi: 10.7326/0003-4819-120-10-199405150-00001. PMID 8154641
- [Background] Freda PU, Beckers AM, Katznelson L, Molitch ME, Montori VM, Post KD, Vance ML; Endocrine Society. Pituitary incidentaloma: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2011 Apr;96(4):894-904. doi: 10.1210/jc.2010-1048. PMID 21474686
- [Background] Rotenberg B, Tam S, Ryu WH, Duggal N. Microscopic versus endoscopic pituitary surgery: a systematic review. Laryngoscope. 2010 Jul;120(7):1292-7. doi: 10.1002/lary.20949. PMID 20578228
- [Background] DeKlotz TR, Chia SH, Lu W, Makambi KH, Aulisi E, Deeb Z. Meta-analysis of endoscopic versus sublabial pituitary surgery. Laryngoscope. 2012 Mar;122(3):511-8. doi: 10.1002/lary.22479. Epub 2012 Jan 17. PMID 22252670
- [Background] Oosmanally N, Paul JE, Zanation AM, Ewend MG, Senior BA, Ebert CS Jr. Comparative analysis of cost of endoscopic endonasal minimally invasive and sublabial-transseptal approaches to the pituitary. Int Forum Allergy Rhinol. 2011 Jul-Aug;1(4):242-9. doi: 10.1002/alr.20048. Epub 2011 Apr 28. PMID 22287427
- [Background] Graham SM, Iseli TA, Karnell LH, Clinger JD, Hitchon PW, Greenlee JD. Endoscopic approach for pituitary surgery improves rhinologic outcomes. Ann Otol Rhinol Laryngol. 2009 Sep;118(9):630-5. doi: 10.1177/000348940911800905. PMID 19810602
- [Background] Suberman TA, Zanation AM, Ewend MG, Senior BA, Ebert CS Jr. Sinonasal quality-of-life before and after endoscopic, endonasal, minimally invasive pituitary surgery. Int Forum Allergy Rhinol. 2011 May-Jun;1(3):161-6. doi: 10.1002/alr.20029. Epub 2011 Apr 26. PMID 22287366
- [Background] Stamm AC, Pignatari S, Vellutini E, Harvey RJ, Nogueira JF Jr. A novel approach allowing binostril work to the sphenoid sinus. Otolaryngol Head Neck Surg. 2008 Apr;138(4):531-2. doi: 10.1016/j.otohns.2007.11.031. No abstract available. PMID 18359368
- [Background] Little AS, Jahnke H, Nakaji P, Milligan J, Chapple K, White WL. The anterior skull base nasal inventory (ASK nasal inventory): a clinical tool for evaluating rhinological outcomes after endonasal surgery for pituitary and cranial base lesions. Pituitary. 2012 Dec;15(4):513-7. doi: 10.1007/s11102-011-0358-4. PMID 22038032
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Wright ED, Agrawal S. Impact of perioperative systemic steroids on surgical outcomes in patients with chronic rhinosinusitis with polyposis: evaluation with the novel Perioperative Sinus Endoscopy (POSE) scoring system. Laryngoscope. 2007 Nov;117(11 Pt 2 Suppl 115):1-28. doi: 10.1097/MLG.0b013e31814842f8. PMID 18075447
- [Background] Doty RL, Shaman P, Dann M. Development of the University of Pennsylvania Smell Identification Test: a standardized microencapsulated test of olfactory function. Physiol Behav. 1984 Mar;32(3):489-502. doi: 10.1016/0031-9384(84)90269-5. PMID 6463130